CLINICAL TRIAL: NCT06687720
Title: A Preliminary Investigation of the Safety and Effectiveness of Oral Probiotics Supplementation for Management of Irritable Bowel Syndrome: A Randomized, Open Label, Placebo-Arm, Comparative, Interventional, Proof-of-Science Study
Brief Title: A Clinical Study to Determine the Safety and Efficacy of An Oral Probiotic Supplementation in the Management of Irritable Bowel Syndrome With Protein Digestion.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Meteoric Biopharmaceuticals Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NB240026-MB
Record Dates: First submitted 2024-11-06; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MetBroma (Experimental): Active Ingredients: Bromelain Mode of Usage: Take one slow-release capsule twice a day, after meal with water Dosage Form: Capsule Unit Dose Route of administration: Oral frequency: Twice a day
  Interventions: Other: MetBroma
- Placebo (Placebo Comparator): Mode of Usage: Take one slow-release capsule twice a day, after meal with water Dosage Form: Capsule Unit Dose Route of administration: Oral frequency: Twice a day
  Interventions: Other: MetBroma

INTERVENTIONS:
Other: MetBroma — Mode of Usage: Take one slow-release capsule twice a day, after meal Dosage Form: Capsule Unit Dose Route of administration: Oral frequency: Twice a day

SUMMARY:
This is an open-label, two-arm, prospective, interventional, in-use safety and efficacy study of an oral probiotic supplementation in adult subjects having irritable bowel syndrome.

DETAILED DESCRIPTION:
A total of the up to 18 adults aged between 18 and 60 years, with irritable bowel syndrome will be enrolled to ensure 16 subjects complete the study.

Subjectsshall be instructed to visit the facility for the following scheduled visits:

* Visit 01 [Within 30 days]: Screening, Blood Parameter Assessment.
* Visit 02 [Day 01]: Enrolment, Evaluations, Treatment Dispensing.
* Visit 03 [Day 15 (±2 days)]: Telephonic follow-up.
* Visit 04 [Day 30 (±2 days)]: Treatment End, Final Evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is an adult male or female aged between 18 to 60 years old.
2. Clinically diagnosed with irritable bowel syndrome (IBS) based on Rome IV criteria: Abdominal pain at least 4 days per month - over at least 2 months - associated with one or more of the following:

   i. Related to defecation ii. A change in frequency of stool iii. A change in form (appearance) of stool iv. After appropriate evaluation, the symptoms cannot be fully explained by another medical condition
3. The subject is having refrigerator at their home for storage of test treatment.
4. The subject is willing to provide written informed consent, comply with the study procedures, and be present for all the visits.
5. The subject is willing to abstain from using any other treatments for irritable bowel syndrome during the study period, unless for a medical urgency.
6. The subject is in a stable medical condition, not requiring immediate intervention or hospitalization.
7. If the subject is female, she is willing to use a highly effective method of contraception throughout the clinical investigation.

   i. Females of childbearing potential must practice and maintain an established method of birth control (e.g., IUD, hormonal implant device/injection, birth control pills, diaphragm, condoms with spermicide, partner vasectomy, or abstinence).

ii. Non-childbearing potential females who are surgically sterile, post-menopausal for at least 1 year, or have had a tubal ligation, must have been using hormonal contraception for at least 6 months and agree to continue using the same contraception for the study duration.

Exclusion Criteria:

1. The subject has a history of diagnosis of either hypertension, diabetes, or liver disease.
2. The subject has any other significant medical condition that could interfere with the study or pose a risk to the participant.
3. The subject has used medications that could influence the study outcomes, such as antibiotics, immunosuppressive drugs, and probiotics or prebiotics supplements within the last 4 weeks.
4. The subject works in frequent night shifts (working night shifts at least 3 times per week), and refuses to change the lifestyle.
5. The subject has a history of alcohol abuse.
6. The subject is either pregnant, lactating, or plans on conceiving during the course of the study.
7. The subject has participated in other clinical studies or received any investigational agent in the previous 30 days.
8. The subject has other significant gastrointestinal diseases (e.g., Crohn's disease, ulcerative colitis, celiac disease).
9. The subject has any condition that, in the investigator's judgment, would compromise the subject's safety or study integrity.
10. The subject has abnormal baseline Haemoglobin (Hb), Complete Blood Count (CBC), Urine Routine/Microscopy (R/M), or Stool Routine/Microscopy (R/M) results that suggest a different pathology than irritable bowel syndrome.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
change in Albumin/Globulin ratio | Baseline before and 6-8 hours post-dose on Day 01 and Day 30
  Evaluate the effect of the test treatment in terms of change in Albumin/Globulin ratio
change in total serum protein | Baseline before and 6-8 hours post-dose on Day 01 and Day 30
  Evaluate the effect of the test treatment in terms of change in total serum protein
change in prealbumin levels | Baseline before and 6-8 hours post-dose on Day 01 and Day 30
  Evaluate the effect of the test treatment in terms of change in prealbumin levels.
Change in the lifestyle using the Scoring and Gradation | Day 01 (before administration) for baseline, and post-dose on Day 30.
  Assessment of the effectiveness of the test treatment in terms of change in the lifestyle using the Scoring and Gradation.
  Severely disturbed lifestyle- 76%-100% Marked disturbed lifestyle-51%-75% Moderately disturbed lifestyle -25%-50% Mild disturbed lifestyle<25
Scoring and Gradation of symptoms of irritable bowel syndrome | Day 01 (before administration) for baseline, and post-dose on Day 30.
  Evaluate of the effect of test treatment using Scoring and Gradation of symptoms of irritable bowel syndrome.
  Complete remission-76%-100% Marked improvement-51%-75% Mild improvement-25%-50% Unchanged<25%

SECONDARY OUTCOMES:
Performance of safety laboratory tests including Complete Blood Count (CBC) | on Day 30
  Evaluate the safety of test treatment through the performance of safety laboratory tests including Complete Blood Count (CBC)
Performance of safety laboratory tests including Biochemical tests | on Day 30
  Evaluate the safety of test treatment through the performance of safety laboratory tests including Biochemical tests
Performance of safety laboratory tests including Urinalysis | on Day 30
  Evaluate the safety of test treatment through the performance of safety laboratory tests including Urinalysis
Assessment of the effectiveness of the test treatment in terms of change in CRP levels | on Day 01 (before administration) for baseline, and post-dose on Day 30 (±2 days).
  CRP will be evaluated by Lab Parameters
Assessment of the effectiveness of the test treatment in terms of change in IL-6 levels | On Day 01 (before administration) for baseline, and post-dose on Day 30 (±2 days).
  IL-6 will be evaluated by Lab Parameters

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd

IPD SHARING:
Plan to Share IPD: No